CLINICAL TRIAL: NCT03425448
Title: Neutrolin Versus Heparin for Locking Hemodialysis Catheters: A Multi-center, Double-Blind, Randomized Controlled Trial
Brief Title: Neutrolin Versus Heparin for Locking Hemodialysis Catheters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Principal Investigator, Dr. Mubarak Al Abdalla, Consultant Nephrologist and Assistant Professor, King Abdullah International Medical Research Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RC17/083/R
Record Dates: First submitted 2018-01-25; First posted 2018-02-07 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Hemodialysis Catheter Infection; Catheter Thrombosis
MeSH Terms: interventions — Heparin

STUDY DESIGN:
Intervention Model Description: Multi-center, double-blind, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heparin group (Active Comparator)
  Interventions: Drug: Heparin
- Neotrolin Group (Experimental)
  Interventions: Device: Neutrolin

INTERVENTIONS:
Drug: Heparin — Heparin hemodialysis catheter lock solution
  Arms: Heparin group
Device: Neutrolin — Neutrolin hemodialysis catheter lock
  Arms: Neotrolin Group

SUMMARY:
Hemodialysis catheter related bacterial infections represent a major cause of mortality and morbidity in the hemodialysis population. Several locking agents had been tried with variable degree of success but not without side effects.

Neutrolin catheter locking agent comprises of heparin,citrate and trauolidine that had been studied in a prospective study in Germany, and it demonstrated a very good result in terms of reducing the catheter related infections and thrombosis.

This study is a multi-center, double-blind RCT comparing the hemodialysis catheter locking solution Neutrolin with heparin in reducing the rate of catheter related bacterial infection and thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* New hemodialysis catheter
* Subject who will need chronic hemodialysis at least twice/week
* Subject likely to require for at least 120 days
* Subject or relative is likely to understand the nature of the study and sign the consent
* Age 18 years and older

Exclusion Criteria:

* Subject with unstable malignancy
* Subject with liver cirrhosis with encephalopathy
* Subject know to have allergy to heparin, citrate or traoulidine
* Documented history of arterial thrombosis or known to have hypercoagulable state
* Subjects with active skin infections and ulcers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2019-04-04 (Estimated); Primary Completion 2020-10-04 (Estimated); Study Completion 2021-04-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of catheter related blood stream infections (CRBSI per 1000 CVC days) | 18 month
  Rate of hemodialysis catheter in each study arm

SECONDARY OUTCOMES:
Proportion of hemodialysis catheters with poor flow due to thrombosis | 18 month
  Rate of catheter dysfunction in each group

IPD SHARING:
Plan to Share IPD: No